CLINICAL TRIAL: NCT07326722
Title: Delivering Transcutaneous Auricular Neurostimulation to Reduce Heavy Menstrual Bleeding: The LUNA Study
Brief Title: Delivering tAN to Reduce HMB: The LUNA Study
Acronym: LUNA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: Lindus Health (Industry); Wellcome Leap (Unknown); Oregon Health and Science University (Other); University of Michigan Health (Unknown); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5L-BLD-06
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Heavy Menstrual Bleeding
Keywords: transcutaneous auricular neurostimulation; tAN; heavy menstrual bleeding; HMB; adolescent heavy menstrual bleeding; aHMB; neurostimulation; vagus nerve stimulation; hemostasis; menstruation; menstrual cycle; blood loss; PBAC; Menorrhagia
MeSH Terms: conditions — Menorrhagia; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two stimulation groups (active tAN or sham tAN) in a 1:1 fashion such that each group will have 20 adult participants and 20 adolescent participants with complete data.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tAN (Experimental): In the Treatment Phase (M3-M5), participants will self-administer one two-hour session of active transcutaneous auricular neurostimulation (tAN) each day of menstruation.
  Interventions: Device: Sparrow Link
- Sham tAN (Sham Comparator): In the Treatment Phase (M3-M5), participants will self-administer one two-hour session of sham transcutaneous auricular neurostimulation (tAN) each day of menstruation. Participants in the sham group will apply the earpiece and connect the cable to the Patient Controller. The device will be turned on, and appears to function identically to an active device, but will not deliver stimulation through the earpiece.
  Interventions: Device: Sparrow Link (Sham)

INTERVENTIONS:
Device: Sparrow Link — The Sparrow Link will be using the components of the Sparrow Ascent device: (FDA-cleared K230796) a wearable, battery-operated, neurostimulation system designed to transcutaneously stimulate nerves on and/or around the auricle.
  Other Names: Transcutaneous Auricular Neurostimulation
  Arms: Active tAN
Device: Sparrow Link (Sham) — Participants will have the earpiece applied and the cable connected to the Patient Controller, but tAN stimulation will not be turned on. The sham device has an identical appearance to the active device.
  Other Names: Transcutaneous Auricular Neurostimulation (Sham)
  Arms: Sham tAN

SUMMARY:
The LUNA study is a prospective, randomized, double-blind, sham-controlled, decentralized clinical trial in participants with heavy menstrual bleeding of no known structural cause. The study includes two age-based cohorts: adolescents aged 14-21 and adults aged 22-45. Participants in both cohorts will be randomized to receive transcutaneous auricular neurostimulation (tAN), which targets the auricular branch of the vagus nerve (ABVN) and the auriculotemporal nerve (ATN), or sham stimulation. Participants will be enrolled into the study over the course of five consecutive menstrual cycles. All study activities will occur remotely and in addition to participants' typical treatment for HMB (as allowed by the eligibility criteria).

During the first two consecutive menstrual cycles (M1 - M2, "Baseline Phase"), no tAN treatment will be delivered. Participants will estimate blood loss using the Pictorial Bleeding Assessment Chart (PBAC), and menstrual cramp pain will be assessed with a Numerical Rating Scale (NRS), daily throughout the duration of the menstruation phase of their two baseline menstrual cycles. Menstrual symptoms will be assessed using the Cox Menstrual Symptom Scale (CMSS) and a general quality of life assessment will be conducted on the final day of menstruation using the RAND Short-Form 36 (RAND-36). Menstrual-related quality of life assessments will also be conducted on the final day of each menstruation using the Menstrual Bleeding Questionnaire (MBQ) in the adult cohort, and the adolescent version (aMBQ) in the adolescent cohort.

During the following three consecutive menstruations (M3 - M5, "Treatment Phase"), participants will self-administer one 2-hour sham or active tAN session daily, beginning Day 1 of menstruation through the final day of menstruation in each menstrual cycle. Blood loss (via the PBAC) and menstrual cramp pain (via the NRS) will be assessed daily throughout the duration of each menstruation. Quality of life will be assessed with the CMSS, RAND-36, and the MBQ (adults) or aMBQ (adolescents) on the final day of each menstruation. A device usability survey will be completed at the end of M3 and M5. Participants will exit the study after the final day of M5.

ELIGIBILITY:
Inclusion Criteria:

1. Regularly menstruating female aged 14-45 years at time of screening
2. History of menorrhagia as assessed by the Menorrhagia Screening Tool
3. Stable/consistent use of current non-hormonal medications and supplements for the past three months, willingness to continue use for duration of study, and not start any new medications or homeopathic remedies
4. Reliable access to an internet-enabled device to complete required questionnaires that is compatible with the study application (iOS 18 and Android 15 or greater)
5. Willingness to consistently use only study-provided menstrual products throughout duration of the study
6. Participant PBAC scores are ≥150 for both baseline menstruation months

Exclusion Criteria:

1. Pregnancy within three months of enrollment
2. Lactating at the time of enrollment
3. Typical length of menstruation greater than 14 days
4. Antifibrinolytic (i.e. tranexamic acid; Lysteda) use within 14 days of enrollment
5. Known acquired bleeding disorder
6. Known severe bleeding disorder (participants with mild von Willebrand disease will be eligible to participate in the study)
7. Use of anticoagulants (i.e. Warfarin, Coumadin, etc.) including platelet inhibitors for 14 days prior to enrollment
8. Use of prescriptive pain medications and/or use of the following analgesics: Aspirin, naproxen (Aleve), or magnesium salicylate (Doan's) during the study
9. Use of the copper intrauterine device within the past three months
10. Structural cause of heavy menstrual bleeding (e.g. fibroids, polyps, etc.) in medical records
11. Thrombocytopenia within the last 12 months (platelet count ≤100,000 per microliter of blood) in medical records
12. Any use of continuous hormone therapies (e.g., IUD, etc.) within three months prior to enrollment
13. Use of hormone therapies that have not followed a standard 21/7 dosing regimen for at least six months prior to enrollment
14. Participant has a history of chronic tobacco use or has ingested nicotine via smoking, vaping, smokeless tobacco, or nicotine patches in the past three months
15. Participant has a history of epileptic seizures within the past 12 months
16. Participant has a history of neurologic diseases (i.e. stroke, brain tumor, cerebrovascular, etc.)
17. Participant has a history traumatic brain injury within the past 12 months
18. Participant has had a splenectomy
19. Participant has presence of devices (e.g., pacemakers, cochlear prostheses, neurostimulators) and/or uses other neurostimulators
20. Participant has abnormal ear anatomy or ear infection present
21. Participant has previously used auricular neurostimulation for any clinical indication
22. Participant is currently or plans to be enrolled in another clinical trial during enrollment
23. Participant is a ward of the state
24. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Regularly menstruating females.
Enrollment: 80 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Pictorial Bleeding Assessment Chart (PBAC) | Daily throughout all five menstruations (up to 5 complete menstrual cycles - estimated 150 days)
  The PBAC is a widely accepted tool for patients with HMB to account for menstrual blood loss. Menstrual blood loss is estimated through a selection of images of tampons, pads, clots, and flooding events. Users mark a tally next to the images that best match each the saturation level of the menstruation products they used that day. PBAC data will be recorded by the participants for each calendar day (00:00-23:59 local time). Day 1 is the calendar date on which a menstrual product is first used. This trial will utilize a modified version of the Higham PBAC, where a tally system will be added to each of the images.

SECONDARY OUTCOMES:
Cox Menstrual Symptom Severity Scale (CMSS) | Final day of each menstruation (up to 5 complete menstrual cycles - estimated 150 days)
  The CMSS measures menstrual distress and dysmenorrhea. The CMSS Severity subscale is an 18-item self-reported scale that measures severity of menstrual symptoms, including pain, nausea, emotions, etc. during menstruation. The CMSS will be used in this trial to retrospectively measure the frequency and severity of a participant's menstrual symptoms on the final day of each menstruation.
Numerical Rating Scale (NRS) | Daily throughout all five menstruations (up to 5 complete menstrual cycles - estimated 150 days)
  The NRS measures menstrual pain daily on a scale of 0 to 10, with zero representing no pain and 10 representing the worst pain imaginable. This is a commonly used scale in studies of dysmenorrhea and other gynecological pain conditions. The NRS will be used in this trial to measure the severity of a participant's menstrual pain on each day of each menstruation.
RAND Short Form-36 (RAND-36) | Final day of each menstruation (up to 5 complete menstrual cycles - estimated 150 days)
  The RAND-36 is a 36-item patient-reported questionnaire that assesses general quality of life. This questionnaire includes eight variables: physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy and vitality, pain, and general perception of health. This questionnaire will be completed by the participant at the end of each menstruation.
Menstrual Bleeding Questionnaire (MBQ) | Final day of each menstruation (up to 5 complete menstrual cycles - estimated 150 days)
  The MBQ measures the impact of heavy menstrual bleeding on health-related quality of life in adult women. The MBQ is a 20-item self-reported scale that evaluates the frequency and severity of menstrual symptoms and their effects on physical, social, and emotional functioning, daily activities, and overall well-being. Responses are captured on Likert-type scales, with higher scores indicating greater symptom burden and functional impairment. The MBQ will be used in this trial to measure the severity of the adult cohort's menstrual pain on the final day of each menstruation.
Adolescent Menstrual Bleeding Questionnaire (aMBQ) | Final day of each menstruation (up to 5 complete menstrual cycles - estimated 150 days)
  The aMBQ measures HMB-related quality of life in adolescents. The aMBQ is a 19-item self-reported scale that evaluates symptom burden and its effects on school attendance and performance, extracurricular and social activities, physical functioning, and emotional well-being, using Likert-type responses with higher scores indicating greater impact. The aMBQ will be used in this trial to measure the severity of the adolescent cohort's menstrual pain on the final day of each menstruation.
Device Usability Questionnaire | Final day of Menstruation 3 and Menstruation 5 (estimated 10 days per menstruation)
  The Device Usability Questionnaire is a 16-item survey that includes both Likert-scale questions (ranging from Strongly Agree to Strongly Disagree) and open-ended free-text responses. It is designed to assess participants' overall satisfaction with the device and to evaluate how easily they were able to operate it using the provided instructions and support materials (Instruction for Use and Quick Start Guide).

CONTACTS AND LOCATIONS:
Overall Officials: Navid Khodaparast, PhD, Principal Investigator — Spark Biomedical, Inc.
Locations (1):
- Lindus Health - DECENTRALIZED STUDY, Boston, Massachusetts, United States